CLINICAL TRIAL: NCT02033252
Title: Acupuncture for Persistent Allergic Rhinitis Complicated With Asthma, A Randomized Controlled Pilot Trial
Brief Title: Acupuncture for Rhinitis Complicated With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun-Yong Choi (Other)
Responsible Party: Sponsor-Investigator, Jun-Yong Choi, Assistant Professor, Korean Medicine Hospital of Pusan National University
Organization: Korean Medicine Hospital of Pusan National University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCRC-KIM-02
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Asthma | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Acupuncture (Experimental): A series of acupuncture sessions within four weeks from the baseline with concurrent conventional medications for asthma
  Interventions: Device: Acupuncture
- Waiting (No Intervention): Participants who will be allocated to waitlist will receive no acupuncture treatments throughout the 4 weeks while receiving other conventional managements for asthma. After 4 weeks, if participants choose to try the acupuncture treatment, the active acupuncture treatment will be provided for 4 weeks (3 sessions/week).

INTERVENTIONS:
Device: Acupuncture — In the acupuncture treatment group, 10 acupuncture points (bilateral LI4, TE23, ST36, unilateral EHN-1, GV23, LI20 and LI4) will be inserted with 0.20 mm in diameter x 30 mm in length disposal needles. The needle will be inserted to a depth of 10 - 30 mm, according to the points selected. The participating acupuncture doctors will manually manipulate the acupuncture needles with de-qi sensation and maintain the needles for 10 minutes with two times of manual stimulation, at the beginning and at the end.
  Arms: Acupuncture

SUMMARY:
This randomized controlled study aimed to evaluate the efficacy and safety of acupuncture therapy on persistent allergic rhinitis patients complicated with asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Suffering from persistent Allergic rhinitis (PAR; nasal obstruction, rhinorrhoea, sneezing and nasal itching) symptoms for more than 4 days/week, and greater than 4 consecutive weeks.
2. Moderate-severe symptoms according to Allergic rhinitis and its impact on asthma (ARIA) criteria.
3. Positive reaction for more than or equal to one respiratory allergen (SPT or MAST)
4. Stable asthma symptoms with diagnosis of Asthma by respiratory or allergic disease specialist.
5. No changes in asthma or allergic rhinitis drugs for the past month
6. Aged greater than or equal to 18 years, either sex.
7. No problem with expression of opinion
8. Provided with written consent
9. No other disease except allergic rhinitis or asthma which could affect the disease.

Exclusion Criteria:

1. Having experience using ventilator due to exacerbation of asthma symptoms within six months.
2. Experience of acute respiratory tract infection treated with antibiotics within 14 days
3. Having anatomical occlusion or deformation in nasal cavity.
4. Signs of infection in chest X-ray or having active respiratory disease except asthma
5. Below or equal to 4 on Total nasal symptom score (TNSS) in the latest week.
6. Received drugs affecting directly to allergic rhinitis such as H1-antihistamines, decongestants (nasal, oral or ocular), corticosteroids within 14 days.
7. Received following treatments for allergic rhinitis or asthma within six months ; Traditional Korean medicine interventions such as acupuncture, moxibustion, cupping therapy and herbal medication inhalation or CAM including homeopathy.
8. Received herbal medication for allergic rhinitis or asthma within 14 days.
9. Pregnant, planning the pregnancy or breast-feeding
10. Tuberculosis, hepatitis or more than 2 x normal limit of serum creatinine, aspartate aminotransferase/alanine aminotransferase (AST/ALT).
11. Skin lesion on acupoint or other systemic disease insufficient for acupuncture.
12. Night-shift workers staying up all night
13. Who cannot participate clinical trial properly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Change from Baseline TNSS Score at 4 Weeks after Randomization

SECONDARY OUTCOMES:
Rhinitis Quality of Life Questionnaire (RQLQ) | Change from Baseline at 2 Weeks after Randomization (Both Groups), Change from Baseline at 4 Weeks after Randomization (Both Groups), Change from Baseline at 8 Weeks after Randomization (Active Group Only)
Quality of Life Questionnaire for adult Korean Asthmatics (QLQAKA) | Change from Baseline at 2 Weeks after Randomization (Both Groups), Change from Baseline at 4 Weeks after Randomization (Both Groups), Change from Baseline at 8 Weeks after Randomization (Active Group Only)
Visual Analogue Scale | Change from Baseline at 2 Weeks after Randomization (Both Groups), Change from Baseline at 4 Weeks after Randomization (Both Groups), Change from Baseline at 8 Weeks after Randomization (Active Group Only)
Pulmonary function test (PFT) | Baseline, four weeks after randomization (both groups)
Euro Quality of Life-5 Dimention Questionnaire (EQ-5D) | Baseline, four weeks after randomization
Total Nasal Symptom Score (TNSS) | Change from Baseline at 2 Weeks after Randomization (Both Groups), Change from Baseline at 8 Weeks after Randomization (Active Group Only)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Yong Choi, KMD, PhD, Principal Investigator — Korean Medicine Hospital, Pusan National University; Yun Seong Kim, MD, PhD, Principal Investigator — Yangsan Pusan National University Hospital; Seung Eun Lee, MD, Study Director — Yangsan Pusan National University Hospital
Locations (1):
- National Clinical Research Center, Korean Medicine Hospital, Pusan National University, Yangsan, Kyungsangnamdo, South Korea